CLINICAL TRIAL: NCT04670146
Title: Prospective Analysis of Epidemiological, Anatomical and Surgical Aspects Leading to a Limitation of the Opening of the Mouth Before and After Oral Cancer Surgery
Brief Title: Understanding Non-radiotherapy-based Development of Trismus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Maximiliaan Smeets, Main investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S63300
Record Dates: First submitted 2020-11-12; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Trismus; Oral Cancer
MeSH Terms: conditions — Trismus; Mouth Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound of the masseteric muscle — Ultrasound of the masseteric muscle to evaluate the thickness and rigidity of the masseteric muscle before and after oral cancer treatment. There will be no invasive investigation of the muscle.

SUMMARY:
A limited mouth opening (or trismus) after surgery for oral cancers is not only one of the most common complications, but it is also a major contributing factor towards an impaired quality of life after surgery. The enormous impact on the quality of life is secondary to impeded speech, feeding, drinking, and aesthetics.

The aim would be to analyse the opening of the mouth before and after surgery, and if applicable after radiotherapy, in a prospective way in oral cancer cases. There is namely a major discrepancy in current science research between the effect of different treatment modalities on trismus, as, in contrast with known research regarding the effect of surgery on trismus, a clear relation between radiotherapy and trismus has already been demonstrated in multiple research articles and systematic reviews. Nevertheless, the clinical experience of this research group supports the need for further investigation on the impact of surgery and the different modalities of surgery on trismus.

The investigators are convinced that revealing the surgical factors, linked with trismus, can lead to better prevention and prediction of later trismus for newly diagnosed oral cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a newly diagnosed oral cancer.
* Cases with a limited mouth opening secondary to oral tumour resections

Exclusion Criteria:

* Minors.
* Deceased cases within the follow-up period of one year.
* Other malignancies than oral squamous cell carcinomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The evaluation of the maximal mouth opening. | Follow-up of twelve months.
  A first endpoint would be to compare the effect of the epidemiological and surgical variables on the maximal mouth opening in millimeters over time.
A detailed quality of life assessment. | Follow-up of twelve months.
  This research group would like to obtain a detailed image of the impact of trismus and oral cancer resections in general on the quality of life. Results will be based on validated and commonly used questionnaires addressing the different aspects of quality of life for this specific population. More specific the Washington questionnaire.
The correlation between the muscles of mastication and trismus. | Follow-up of twelve months.
  Investigation of the relation between the muscles of mastication and the tumour and how this correlation influences the incidence of postsurgical trismus. Therefore, the distance between the tumor and the muscles of mastication will be evaluated in millimeters, based on 3D preoperative radiological imaging (CT or MRI).
An evaluation of the masseter muscle via ultrasound before and after oral tumor resections/trismus treatment. | Follow-up of twelve months.
  The final endpoint will be the evaluation of masseter alterations on ultrasound, which will lead to an improved understanding of muscular changes due to oncological resections, radiotherapy, and trismus. Even though newer (IMRT or intensity-modulated radiation therapy) techniques in radiotherapy protect vital structures as much as possible, the masseter is still often involved in the radiated area and muscular alterations are anyhow to be expected. The endpoints will be alterations in masseter muscle thickness (millimeter) in all oral oncology cases, trismus patients secondary to oral oncology resections, and in adjuvant radiotherapy cases.
Correlation of the mouth opening with surgical variables. | Follow-up of twelve months.
  The use of free vascularized grafts (primary closure/skin graft/composite grafts/soft tissue free flaps) and a neck dissection (yes/no) will be analyzed to identify an impact on the mouth opening of each surgical variable to prevent trismus in future cases. The information will be collected from the electronic patient file.
Correlation of the mouth opening with tumor stage. | Follow-up of twelve months.
  The correlation between tumor stage(I-IV) (TNM-classification according to TNM-8 AJCC manual) and mouth opening will be analyzed. The information will be collected from the electronic patient file.
Correlation of the mouth opening with tumor recurrence. | Follow-up of twelve months.
  An evaluation of the influence of tumor recurrence (yes/no) on the maximal mouth opening will be ordered. The information will be collected from the electronic patient file.
A detailed quality of life assessment regarding head and neck cancer treatment. | Follow-up of twelve months.
  This research group would like to obtain a detailed image of the impact of trismus and oral cancer resections in general on the quality of life. Results will be based on validated and commonly used questionnaires addressing the different aspects of quality of life for this specific population. More specific the EORTC H&N 35.
A detailed quality of life assessment regarding the mouth opening. | Follow-up of twelve months.
  This research group would like to obtain a detailed image of the impact of trismus and oral cancer resections in general on the quality of life. Results will be based on validated and commonly used questionnaires addressing the different aspects of quality of life for this specific population. More specific the Gothenburg questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bila, MD, DDS, Principal Investigator — KU Leuven
Locations (1):
- Omfs-Impath, Leuven, Vlaams-Brabantt, Belgium

IPD SHARING:
Plan to Share IPD: Yes